CLINICAL TRIAL: NCT01890161
Title: A Phase IIa Randomized Double-blind Placebo-controlled Two-way Cross-over Trial of the Effects of Repeat Doses of 50 mg AXP1275 Daily on the Asthmatic Response to a Pulmonary Allergen Challenge in Adults With Mild-to-Moderate Atopic Asthma
Brief Title: A Phase IIa Repeat Dose AXP1275 vs Placebo Cross-over Trial With Pulmonary Allergen Challenge in Adults With Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Axikin Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AXP1275-201
Record Dates: First submitted 2013-06-26; First posted 2013-07-01 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-01

CONDITIONS: Atopic Asthma
Keywords: asthma
MeSH Terms: conditions — Asthma | interventions — AXP1275

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AXP1275 (Experimental): AXP1275 50 mg (2 × 25-mg capsules) once daily for 14 days
  Interventions: Drug: AXP1275
- AXP1275 matching placebo (Placebo Comparator): AXP1275 matching placebo (2 capsules) once daily for 14 days
  Interventions: Drug: AXP1275 matching placebo

INTERVENTIONS:
Drug: AXP1275 — AXP1275 50 mg (2 × 25-mg capsules)
  Arms: AXP1275
Drug: AXP1275 matching placebo — AXP1275 matching placebo (2 capsules)
  Arms: AXP1275 matching placebo

SUMMARY:
This is the first study in human patients with asthma that the sponsor is conducting in order to evaluate if there are signals that the investigational medication, AXP1275, may be a safe and effective treatment for asthma. The results of this study may help the sponsor to design additional studies.

DETAILED DESCRIPTION:
This 2-way, randomized, double-blind crossover study in subjects with mild to moderate atopic asthma is designed to compare the responses to allergen and methacholine challenges within the same subject after approximately 2 weeks of treatment with AXP1275 50 mg or placebo. A total of 20 subjects with asthma with a dual (early and late) asthmatic response to an inhaled aeroallergen will be randomized to 1 of 2 treatment sequences (placebo then AXP1275 or AXP1275 then placebo) in a double-blind fashion to receive either oral AXP1275 or matching placebo, once-daily, for 14 days. The washout period between the 2 treatment periods will be 14 to 21 days.

A post-treatment follow-up visit will occur 14 ± 3 days after completion of the second treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 64 years (inclusive).
2. Male or female.
3. If male, is surgically sterile (vasectomy) or agrees to comply with required contraceptive measures.
4. If female, not pregnant (or lactating), as evidenced by a negative serum pregnancy test, and is either surgically sterile (hysterectomy, bilateral ovariectomy, or bilateral tubal ligation), or if a female of childbearing potential, agrees to comply with required contraceptive measures.
5. History of episodic wheeze and shortness of breath with a prebronchodilator FEV1 ≥70% of predicted at screening.
6. Asthma symptoms treated (if necessary) only with intermittent short-acting ß-agonist therapy by inhalation.
7. Demonstration of a positive wheal reaction on skin prick testing to at least 1 common aeroallergen at screening.
8. Screening inhalational allergen challenge response demonstrating that the subject experiences both an early asthmatic response (EAR) and a late asthmatic response (LAR).
9. Methacholine PC20 ≤16 mg/mL at screening.
10. No history of smoking within 6 months of screening, and with a total pack year history of ≤10 pack years.
11. 12-lead ECG recording without signs of clinically relevant pathology or showing no clinically relevant deviations as judged by the investigator.
12. All values for hematology, clinical chemistry, and urinalysis within the normal range, or if abnormal, are deemed not clinically significant by the investigator with documented agreement from the medical monitor.
13. Is able to give written informed consent.

Exclusion Criteria:

1. Past or present disease which, as judged by the investigator, may affect the outcome of this study.
2. Respiratory tract infection and/or exacerbation of asthma within 4 weeks prior to the screening period.
3. Symptomatic allergic rhinitis. Those subjects with a history of allergic rhinitis may participate if asymptomatic at screening (and continue to be so at baseline on Day 1 prior to dosing) and if, in the opinion of the investigator, it is unlikely that disease exacerbation will occur during the course of the study.
4. History of life-threatening asthma.
5. Abnormal chest X-ray.
6. Use of oral, injectable, or dermal steroids within 3 months and/or inhaled steroids within 1 month of screening.
7. Use of cromoglycate, nedocromil, leukotriene receptor antagonists (zafirlukast, pranlukast, montelukast), and inhibitors of 5-lipoxygenase (zileuton) within 4 weeks of screening.
8. Use of immunosuppressives, anticoagulants (warfarin or heparin), or any medications that may interact with pharmacodynamic (PD) effects of AXP1275 within 4 weeks of screening.
9. Use of theophylline-containing agents (any type) and long-acting β2-agonists (salmeterol, formoterol) within 4 weeks of screening.
10. Positive screen for drug(s) of abuse (opiates, methadone, cocaine, amphetamines, cannabinoids, barbiturates, or benzodiazepines) or cotinine.
11. Positive for hepatitis B surface antigen, hepatitis C virus, or human immunodeficiency virus (HIV) 1/2.
12. Has participated in a clinical trial and has received an investigational product within 30 days prior to screening, or 5 elimination half lives of the investigational product, whichever is longer.
13. Has had significant blood loss (>500 mL) or donation of blood within 2 months prior to screening visit 1.
14. History of being unable to tolerate or complete methacholine or allergen challenge tests.
15. Subject is undergoing allergen desensitization therapy.
16. History of immunotherapy in the 3 years prior to screening or concurrently undergoing immunotherapy treatment.
17. Professional or ancillary personnel involved in the study.
18. Is not, in the opinion of the investigator, suitable for entry into the study.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2013-08; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Late Asthmatic Response | From 3 to 7 hours after allergen challenge on day 13 of both 14-day treatment periods
  Area under the forced expiratory volume in 1 second (FEV1) curve from 3 to 7 hours after allergen challenge (AUC3-7h) on day 13 of both 14-day treatment periods.

SECONDARY OUTCOMES:
Early Asthmatic Response | Between 0 to 2 hours after allergen challenge on day 13 of both 14-day treatment periods
  Maximum percentage fall in FEV1 and AUC of FEV1 between 0 to 2 hours (AUC0-2h) after allergen challenge on day 13 of both 14-day treatment periods.
Late Asthmatic Response-Secondary | Between 3 to 7 hours after allergen challenge on day 13 of both 14-day treatment periods
  Maximum percentage fall in FEV1 between 3 to 7 hours after allergen challenge on day 13 of both 14-day treatment periods.
Total Asthmatic Response | Between 0 to 7 hours after allergen challenge on day 13 of both 14-day treatment periods
  Minimum FEV1 and AUC of FEV1 between 0-7 hours (AUC0 7h) after allergen challenge on day 13 of both 14-day treatment periods.
FEV1 comparison | At day 12, 13, and 14 of both 14-day treatment periods
  For FEV1 values at each time point on day 12, 13, and 14, the difference between the two treatments will be calculated.
Sputum eosinophil count | On days 12, 13, and 14 of both 14-day treatment periods
  Induced sputum eosinophil count per mL of sputum on days 12, 13, and 14 of both 14-day treatment periods.
Sputum cell count (other) | On days 1, 12, 13, and 14 of both 14-day treatment periods
  Induced sputum cell count per mL of sputum for cells other than eosinophils (including basophils) on days 1, 12, 13, and 14 of both 14-day treatment periods.
CCL13 and CCL17 concentrations | On days 12, 13, and 14 of both 14-day treatment periods
  Comparison of the two treatments for changes in sputum concentrations of CCL13 and CCL17.
Provocative concentration of methacholine | Between days 1 and 12 and between days 12 and 14 of both 14-day treatment periods
  Shift in the provocative concentration of methacholine resulting in a 20% reduction in FEV1 (PC20) between days 1 and 12 and between days 12 and 14 of both 14-day treatment periods.
Maximum exhaled nitric oxide (eNO) and AUC of eNO | On days 13 and 14 of both 14-day treatment periods
  Maximum eNO and AUC of eNO on days 13 and 14 (AUC0-24h) of both 14-day treatment periods.
eNO comparison | On days 13 and 14 of both 14-day treatment periods
  For eNO values at each time point on day 13, and 14 of both 14-day treatment periods, the difference between the two treatments will be calculated.

OTHER OUTCOMES:
Adverse events (AEs) | Throughout both 14-day treatment periods
  The incidence of treatment-emergent AEs will be summarized by system organ class, preferred term, and maximum severity or strongest relationship to study treatment for both treatments. Serious AEs and AEs leading to early withdrawal from the study will also be listed.
Clinical laboratory, vital signs, physical examination, and ECG changes | Baseline to the end of the study (14 +/- 3 days from the last of two treatments)
  Clinical safety laboratory tests data will be listed by subject and visit with values falling outside the normal range provided in a separate listing. Shifts from abnormally low/normal/abnormally high at baseline to the end of the study will be shown.
  Data on physical examinations, vital signs, and ECGs will be listed.
AXP1275 plasma concentrations | day 6 or 7 (predose), day 12 (3 hr post dose), day 13 (3 and 10 hr post dose), and day 14 (3 hr post dose) for the active treatment arm
  AXP1275 plasma concentrations will be evaluated to determine if steady-state has been reached (minimum concentration [Cmin] on day 6 or 7) and for study drug dosing compliance purposes. In addition, concentrations at other time points will be evaluated relative to individual pharmacodynamic responses associated with a given time point.

CONTACTS AND LOCATIONS:
Overall Officials: Paul O'Byrne, MD, Principal Investigator — McMaster University; Louis-Philippe Boulet, MD, Principal Investigator — IUCPQ, Institut de cardiologie et de pneumologie de l'Hôpital Laval; Mark Fitzgerald, MD, Principal Investigator — University of British Columbia, Vancouver General Hospital
Locations (3):
- Canada (3):
  - Vancouver General Hospital, The Lung Centre, Vancouver, British Columbia
  - McMaster University, Hamilton, Ontario
  - IUCPQ, Institut de cardiologie et de pneumologie de l'Hôpital Laval, Québec, Quebec